CLINICAL TRIAL: NCT05239299
Title: Dissemination of Scientific Findings: Wishes and Realities in the Field of Pediatric Chronic Pain
Brief Title: Treatment Options for Pediatric Chronic Pain: How do we Best Disseminate Our Scientific Findings
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Dissemination Focus Groups
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Chronic Pain
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents with chronic pain
  Interventions: Other: No intervention, observational study
- Parents of adolescents with chronic pain
  Interventions: Other: No intervention, observational study
- Health care professionals who work with adolescents with chronic pain
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study — Focus Group

SUMMARY:
Pediatric chronic pain is a prevalent condition with manifold treatment options. However, knowledge of targeted dissemination of intervention research findings is currently lacking.

The aim of this project is to determine satisfaction with current knowledge transfer from science to clinical practice amongst health care professionals, adolescents with CPP and their parents and to understand what treatment options have been offered to patients in Swiss pain centers Three focus groups, one with health care professionals, one with adolescent patients, and one with their parents, will be conducted to determine how the dissemination of scientific evidence to clinical practice can be improved and what hurdles exists when gathering information about pain interventions. In addition, patients will be asked about the treatment options offered to them and health care professionals about which treatments they routinely prescribe and why.

ELIGIBILITY:
Inclusion Criteria:

Adolescent group:

* Adolescents suffering from chronic pain (i.e., persistent or recurrent pain for three months or more)
* Able to read and speak German

Parent group:

* Parents of an adolescent with chronic pain
* Able to read and speak German

Health care professionals group:

* Health care professional working with adolescents with chronic pain
* Able to read and speak German

Exclusion Criteria:

* no chronic pain or experience with chronic pain

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with chronic pain, one of their parents and health care professionals working with adolescents with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-05-21 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Information seeking behavior | immediattely after the focus group
  Participants' key messages will be reduced to major subjects by means of content analysis. The goal is to understand participants' information seeking behavior with regard to chronic pain and interventions for chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Helen Koechlin, PhD, Principal Investigator — University of Basel
Locations (1):
- Faculty of Psychology, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No